CLINICAL TRIAL: NCT02597270
Title: Mapping Natural Polymorphisms of Hepatitis C Virus NS3/4A Protease and NS5A Region Among Brazilian Chronic Patients (MAPPING)
Brief Title: An Observational/Non-interventional, Study of NS3/4a Protease and NS5A Protein of Hepatitis C Virus in Brazilian Participants With Chronic HCV Infection
Acronym: MAPPING
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR107065; TMC435HPC4012 (Other: Janssen-Cilag Ltd.)
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Hepatitis C Virus
Keywords: Hepatitis C virus
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The total blood volume to be collected will be approximately 15 milliliters (mL) (3 tubes, 5mL each). Fasting is not required. The blood sample collection scheme was designed to collect the minimum number of blood samples that is necessary to accomplish the study objective. Blood samples will be frozen and incinerated 30 days after blood collection at the national central laboratory.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Brazilian participants with Genotype 1 HCV infection treatment naive participants or previously failed to double therapy (Peg-interferon-α and Ribavirin) will be included in the trial and will constitute the trial population.

SUMMARY:
The purpose of this study is to describe the genetic diversity of Hepatitis C virus (HCV) NS3/4a protease and NS5A protein of HCV in participants with chronic disease naive-drug or previously failed to double therapy (Peg-interferon and Ribavirin) and to identify the frequency of natural polymorphisms in HCV NS3/4a protease and NS5A protein that are associated with direct-acting antivirals (DAAs)-resistance.

DETAILED DESCRIPTION:
This is a multicenter, observational/non-interventional, cross-sectional study to describe the genetic diversity of and to identify the natural polymorphisms in HCV NS3/4a protease and NS5A protein of hepatitis C virus in Brazilian participants with chronic HCV infection. Brazilian participants with Genotype 1 HCV infection treatment naive participants or previously failed to double therapy (Peg-interferon-α and Ribavirin) will be included in the trial and will constitute the trial population.

ELIGIBILITY:
Inclusion Criteria:

* Participants mono infected with chronic Hepatitis C infection (genotype 1), including naive patients or previously failed to double therapy (Peg-interferon-α and Ribavirin)
* There is no restriction on fibrosis stage or clinical liver disease
* There is no restriction for comorbidities
* Male or female participants with age >=18 years

Exclusion Criteria:

* Participants failed to triple therapy using protease inhibitors
* Participants with co-infections (i.e. Human immunodeficiency virus, Hepatitis B virus)
* Participants that are not agree to sign the written informed consent
* Participants is taking part in an interventional clinical trial with an investigational agent (i.e. non-commercialized agent) or in an interventional clinical trial sponsored by Johnson & Johnson

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Brazilian participants with Genotype 1 HCV infection treatment naive patients or previously failed to double therapy (Peg-interferon-α and Ribavirin) will be included in the trial.
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2016-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants With HCV NS3/4a Protease and NS5A Protein | Day 1
  After extraction of HCV RNA from collected blood samples, the sequences of the NS3/4A and NS5A genes of HCV will be amplified by reverse transcription polymerase chain reaction (RTPCR) using specific primers for each genomic region. PCR products will be sequenced subsequently by direct sequencing. Detection of natural polymorphisms will be analyzed a comparison of the each sequence with the subtype consensus sequence.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (6):
- Brazil (6):
  - Belém
  - Goiânia
  - Porto Alegre
  - Porto Velho
  - Salvador
  - São Paulo